CLINICAL TRIAL: NCT00176150
Title: Influence of Cholesterol Plasma Levels on Drug Transport in Patients With Anorexia Nervosa
Brief Title: Drug Transport in Patients With Anorexia Nervosa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Other Study IDs: K075
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2003-04

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; multidrug resistance; cholesterol metabolism
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The aim of this study is to investigate whether patients with anorexia nervosa have elevated plasma cholesterol levels and, if elevated plasma cholesterol levels influence drug transport by the ABC-transporter P-gp (P-glycoprotein, MDR 1/ABCB1). We will isolate peripheral blood mononuclear cells (PBMCs) and total RNA from the blood of patients with anorexia nervosa and healthy subjects as control. PBMCs will be used for quantitative cholesterol determination and for measuring the activity of P-gp using a FACS (fluorescence-activated cell sorting) method (rhodamine123 efflux). Total RNA will be used for quantitative expression analysis of P-gp by reverse transcriptase real time PCR.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis anorexia nervosa according to DSM-IV (Diagnostic and Statistical Manual of Mental Disorders. Washington, DC) Refusal to gain weight to or over a minimal normal weight (BMI < 17,5 kg/m²) Fear of gaining weight despite underweight

Exclusion Criteria:

Contraindication for taking blood samples (haemoglobin < 8,5 g/dl) Medication which could influence the lipid metabolism (current and the last two months) Acute or chronic diseases, particularly malign diseases Diseases which could affect the safety of the patients or which could interfere with aims of the study Positive pregnancy test Excessive alcohol consumption (more than 30 g alcohol per day) or alcohol consumption within two days before sampling blood Disability to communicate with the investigator because of linguistic problems or because of a limited mental state

Inclusion criteria for healthy subjects:

Age matched with patients with anorexia nervosa (18 years to 30 years) Well status of health Female Negative pregnancy test No clinical relevant diagnosis, particularly no hyperlipoproteinemias (LDL < 160 mg/dl) BMI > 18,0 kg/m² and < 25 kg/m²

Exclusion criteria for healthy subjects:

Medication which could influence the lipid metabolism (current and two months ago inclusively) Acute or chronic diseases, particularly malign diseases Diseases which could affect the safety of the patients or which could interfere with aims of the study Positive pregnancy test Excessive alcohol consumption (more than 30 g alcohol per day) or alcohol consumption within two days before sampling blood Disability to communicate with the investigator because of linguistic problems or because of a limited mental state

Ages: 15 Years to 30 Years | Sex: Female
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Walter Emil Haefeli, Prof. Dr., Principal Investigator — Department of Internal Medicine VI, Clinical Pharmacology and Pharmacoepidemilogy
Locations (1):
- Department of Internal Medicine VI, Clinical Pharmacology and Pharmacoepidemiology, Heidelberg, Germany